CLINICAL TRIAL: NCT04459104
Title: The Association Between Pain, Nutrition and Glycemic Response in Chronic Low Back Pain and Breast Cancer Survivors: a Cross-over Trial.
Brief Title: Pain, Nutrition and Glycemic Response in Chronic Low Back Pain and Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Malfliet Anneleen, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: B1432020000025
Record Dates: First submitted 2020-06-17; First posted 2020-07-07 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain
Keywords: breast cancer survivors; chronic low back pain; nutrition; diet; glycemic response; fasting glucose level; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- chronic low back patients (Experimental): Participants will be given two beverages, (isomaltulose or sucrose) in a random order (one of each on each of the two test dates).
  Interventions: Other: Low glycemic load; Other: High glycemic load
- breast cancer survivors having chronic pain (Experimental): Participants will be given two beverages, (isomaltulose or sucrose) in a random order (one of each on each of the two test dates).
  Interventions: Other: Low glycemic load; Other: High glycemic load
- healthy pain-free controls (Active Comparator): Participants will be given two beverages, (isomaltulose or sucrose) in a random order (one of each on each of the two test dates).
  Interventions: Other: Low glycemic load; Other: High glycemic load

INTERVENTIONS:
Other: Low glycemic load — Participants will be given test beverages containing 50gr of isomaltulose (low glycemic index = 32). Isomaltulose powder will be dissolved in 250mL water, and participants will be instructed to consume this beverage within 5 minutes. Blood glucose levels will be collected at 15, 30, 45, 60, 90, and 120 minutes after consumption of the beverages. The first two drops of blood will be discarded, the third drop will be used for testing.
Other: High glycemic load — Participants will be given test beverages containing 50gr sucrose (high glycemic index = 65). Sucrose powder will be dissolved in 250mL water, and participants will be instructed to consume this beverage within 5 minutes. Blood glucose levels will be collected at 15, 30, 45, 60, 90, and 120 minutes after consumption of the beverages. The first two drops of blood will be discarded, the third drop will be used for testing.

SUMMARY:
The development of chronic pain is one of the most seen sequelae in the cancer survivor population. Literature reports the presence of pain in approximately 40% of 5-year survivors. Specifically, in breast cancer survivors, chronic pain is estimated to be present in at least 50% of this population. On the other hand, chronic low back pain is one of the leading causes of disability and decrease in quality of life. It has huge economical, psychological and social impacts on individuals, society and health institutions.

Unhealthy dietary behavior is associated with the occurrence, maintenance and management of chronic pain. Also, excessive calorie intake and diets rich in sugar, fat, sodium and caffeine were observed in patients having chronic pain. However, although nutritional factors are suggested as an associated lifestyle factor of chronic pain, limited attention is given to dietary and nutritional factors in relation to chronic pain.

One particular mechanism drawing attention in the link between nutrition and pain are blood glucose levels and the glycemic response. Animal research shows the potential for reduced blood glucose to influence several pathways involved in chronic pain, including decreased oxidative stress, and reduced neuronal excitability. Given the link between blood glucose levels, as well as the evidence for the importance of interpersonal variability in the glycemic response, this glycemic response can also be of interest for chronic pain research. Finding a possible link between both the glycemic response and pain-related outcomes, could give direction to further research focussing on implementing (personalized) nutritional/dietary advise to maintain healthy blood glucose levels in people suffering from chronic pain.

Therefore, this study will provide the first step in this promising line of research, by being the first to look for differences in glycemic response between breast cancer survivors having chronic pain and healthy pain-free controls, and between chronic low back pain patients and healthy pain-free controls.

Secondly, this study will also investigate possible associations between glycemic response, pain-related outcomes, nutrition related outcomes, physical activity, and body composition for breast cancer survivors and chronic low back pain patients separately in comparison with healthy pain-free controls.

DETAILED DESCRIPTION:
Study Design:

This study will be carried out as an experimental, cross-over study, including two pain populations, one control group and two assessment sessions.

At the first session, firstly, all participants will undergo an assessment including pain-related outcomes, nutrition-related outcomes, and measures of physical activity, quality of life, body composition, and fasting blood glucose. Secondly, participants will be given a test beverage (with a high or low glycemic index, randomly decided), after which blood glucose levels will be assessed several times during the next 120 minutes.

At the second session, two days later (washout period), only fasting blood glucose levels will be tested again, after which the study participants will be given the other test beverage, after which blood glucose levels will be monitored once more for 120 minutes. Other outcome measures will not be re-assessed after exposure to the beverages, as we do not expect a direct influence of these test beverages on the outcome variables.

Results will be analysed and published separately for chronic low back pain patients and breast cancer survivors.

Recruitment of participants:

Participants will be recruited via posters and flyers. These posters and flyers will also be distributed to general practitioners, pharmacists, physiotherapists, health insurance companies, etc., who will be asked to alert potential participants to the possibility of study participation. Information and recruitment messages will also be placed on the website and social media platforms of the Pain in Motion research group.

Informed consent:

Prior to participating in the studies, each participant will be asked to read and sign a participant information sheet and a consent form

ELIGIBILITY:
GROUP 1=Chronic Low Back Pain

Inclusion Criteria

* Women between 18 and 65 years old;
* Native Dutch speaker;
* Experiencing chronic nonspecific low back pain (i.e. pain present for at least 3 months, at least 3 days per week);
* No new medication or new treatments started in the 6 weeks prior to or during study participation;
* Non-specific failed back surgery can be included if the operation was anatomically successful and happened at least 3 years ago;
* No physical exertions over 3 Metabolic Equivalent of Task (MET) in the 3 days before the assessments;
* No analgesics/ caffeine/ alcohol/ nicotine 48 hours prior to the assessments

Exclusion Criteria

* People who have any other diagnosed systemic diseases e.g. diabetes mellitus, hypertension, cardiovascular diseases etc;
* Participants who have neuropathic pain according to "Douleur Neuropathique 4 Questionnaire" and the S-LANSS Neuropathic Pain Score;
* Chronic widespread pain diagnosis (like fibromyalgia, chronic fatigue syndrome, whiplash);
* Current pregnancy or pregnant in the past year;
* Specific spinal pathology (e.g., hernia, spinal stenosis, spondylolisthesis, infection, spinal fracture or malignancy)

GROUP 2= Breast Cancer Survivors

Inclusion Criteria

* Female breast cancer survivors with chronic pain (lasting at least 3 months, at least 3 days per week);
* Participants between 18 and 65 years old;
* Native Dutch speaker;
* Active treatment ended at least 3 months ago (i.e. surgery, radiotherapy and chemotherapy; hormone and immune therapy can be going on);
* No analgesics/ caffeine/ alcohol/ nicotine 48 hours prior to the assessments

Exclusion Criteria

* People who have any other systemic disease like hypertension, Type II Diabetes etc;
* Current pregnancy or pregnant in the past year;
* Current active cancer process;
* Tube feeding

GROUP 3= Healthy, Pain-Free Controls

Inclusion Criteria

* Female, healthy and pain-free participants between 18 and 65 years old;
* Native Dutch speaker;
* No analgesics/ caffeine/ alcohol/ nicotine 48 hours prior to the assessments

Exclusion Criteria

* Current pregnancy or pregnant in the past year;
* People who have any other diagnosed systemic diseases e.g. diabetes mellitus, hypertension, cardiovascular diseases;
* Participants who have neuropathic pain according to "Douleur Neuropathique 4 Questionnaire" and the S-LANSS Neuropathic Pain Score;
* Chronic widespread pain diagnosis (like fibromyalgia, chronic fatigue syndrome, whiplash);
* Specific spinal pathology (e.g., hernia, spinal stenosis, spondylolisthesis, infection, spinal fracture or malignancy)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Glycemic response | at the 1st day
  Blood glucose levels will be measured using OneTouch Verio (LifeScan Europe, Johnson & Johnson, Switzerland). Blood glucose levels will be collected at 15, 30, 45, 60, 90, and 120 minutes after consumption of the beverages.
Glycemic response | at the 2nd day
  Blood glucose levels will be measured using OneTouch Verio (LifeScan Europe, Johnson & Johnson, Switzerland). Blood glucose levels will be collected at 15, 30, 45, 60, 90, and 120 minutes after consumption of the beverages.

SECONDARY OUTCOMES:
Brief Pain Inventory | at the 1st day
  The "Brief Pain Inventory" allows to rate the worst pain in the last 24 hours, the least pain in the last 24 hours, the average pain and the pain intensity at the moment of filling out the questionnaire. This tool also assesses the interference of pain with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep via an 11-point numeric rating pain scale, ranging from 0 (no pain) to 10 (worst pain).
Central Sensitization Inventory | at the 1st day
  The "Central Sensitization Inventory" assesses symptoms that can indicate central sensitization mechanisms. It includes two sections, Part A and Part B, which can be used independently from each other. In this study, only Part A will be used, which includes 25 questions scored on a Likert Scale ranging from 0 (i.e. never) to 4 (i.e. always). Summing these scores, a total score between 0 and 100 is obtained. The CSI showed a cut-off of 40 to indicate the possible presence of central sensitization.
Douleur Neuropathique 4 Questionnaire | at the 1st day
  The "Douleur Neuropathique 4 Questionnaire" is a screening tool for neuropathic pain. It consists of four main questions, which all include 10 sub-questions. Each of these subquestions can be answered with YES (1 point) or NO (0 points). Scores which are equal or higher to 4 out of 10 indicate the possible presence of neuropathic problems that underly the pain problem.
Electrical Detection Threshold | at the 1st day
  Electrical detection thresholds will be measured using the Surpass LT stimulator (EMS Biomedical, Korneuburg, Austria) at the bilateral sural nerve, and at the bilateral median nerve (i.e. four test sites). Each stimulus will be a constant current rectangular pulse train consisting of 5 pulses delivered at a frequency of 250 Hertz. Stimulation will start at 0 milli amper and will be gradually increased using steps of 0.5 milli amper until the patient is experiencing a faint sensation.
Electrical PainThreshold | at the 1st day
  Electrical pain thresholds will be measured using the Surpass LT stimulator (EMS Biomedical, Korneuburg, Austria) at the bilateral sural nerve, and at the bilateral median nerve (i.e. four test sites). Each stimulus will be a constant current rectangular pulse train consisting of 5 pulses delivered at a frequency of 250 Hertz. Stimulation will start at 0 milli amper and will be gradually increased using steps of 0.5 milli amper until the stimulus is experienced as painful.
Electrical Temporal Summation | at the 1st day
  Electrical temporal summation will be measured using the Surpass LT stimulator (EMS Biomedical, Korneuburg, Austria). Temporal summation will be assessed by delivering 20 electrical stimuli at the previously determined intensity of the electrical pain threshold. The patient will be asked to give a verbal numeric rating scale score ranging from 0 (= no pain) to 100 (= worst possible pain) at the 1st, the 10th and the 20th stimulus. The outcome measures for temporal summation will be the differences between the 10th and 1st pain score, the 20th and 10th pain score and 20th and 1st pain score.
Electrical Offset Analgesia | at the 1st day
  Electrical offset analgesia will be measured using the Surpass LT stimulator (EMS Biomedical, Korneuburg, Austria). Electrical stimuli will be applied as a train of rectangular pulses delivered by a constant current stimulator. The stimulation intensity will be calculated using the electrical pain threshold. The study participants will be given the painful stimuli into three times intervals and using three intensities; T1 (5 seconds at 150% of Electrical pain threshold), T2 (5 second at 180% of Electrical Pain threshold) and T3 (20 seconds at 150% Electrical pain threshold). Afterwards, participants will undergo a control electrical stimulus which encompasses 30 seconds of constant electrical stimulation at 150% of the Electrical pain threshold. During each application (control trial, T1, T2, and T3) participants need to report their intensity of pain on a visual analogue scale. The scale is anchored by "no pain"(score of 0) and "worst imaginable pain" (score of 100).
Pressure Pain Threshold | at the 1st day
  Pressure pain thresholds measure hyperalgesia by means of a digital pressure algometer (Wagner Instruments, Greenwich) with a 1 centimetre square tip. Pressure will be increased at a rate of 1 kilogram per second. Subjects need to say "stop" when the pressure is experienced as painful.
3 day dietary dairy | at the 1st day
  The diary asks for dietary intake information of two weekdays and one day in the weekend. Collected data with the 3-day food diary will allow us to find out approximate calorie intake, micronutrient intake, macronutrient intake of each participant.
Healthy Eating Index | at the 1 st day
  Collected data with the 3-day food diary will allow us to calculate the Healthy Eating Index. The "Healthy Eating Index" consists of thirteen items of which nine items (total fruit, whole fruit, vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids) are recommended to consume, while the consumption of the other four items (refined grains, sodium, added sugars, saturated fats) should be as low as possible in order to achieve a healthy diet. Score for the Healthy Eating Index range from 0 to 100. Higher scores represent healthier diets
Mediterranean Diet Score | at the 1st day
  A nine-point score of the Mediterranean Diet Score can be calculated using gender-specific medians of intake. A value above the median is rated 1, below the median 0. Higher scores represent healthier diets.
Short Form- 36 Quality of Life | at the 1st day
  "Short Form-36" contains 36 questions across 7 subscales, namely, "general health", "limitations of activities", "physical health problems", "emotional health problems", "social activities", "pain" and "energy and emotions". Each domain ranked between 0 to 100. Higher scores indicates better.
International Physical Activity Questionnaire | at the 1st day
  The "International Physical Activity Questionnaire" consists of 5 main domains (1-job-related physical activity; 2-transportation related physical activity; 3-housework, house maintenance, and caring for family-related physical activity; 4-recreation, sports, and leisure-time physical activity; and 5-time spent sitting) with 27 context-specific physical activity questions. Higher scores indicates better.
Body Weight | at the 1st day
  "TANITA MC-780MA" bio electrical impedance analysis will be used to analyse the body weight in kilograms and body weight percentage.
Body fat mass | at the 1st day
  "TANITA MC-780MA" bio electrical impedance analysis will be used to analyse the body fat mass in kilograms and body fat mass percentage.
Body muscle mass | at the 1st day
  "TANITA MC-780MA" bio electrical impedance analysis will be used to analyse the body muscle mass in kilograms and body muscle mass percentage.
Body water | at the 1st day
  "TANITA MC-780MA" bio electrical impedance analysis will be used to analyse the body water in kilograms and body water percentage.
Body Height | at the 1st day
  Body height in meters will be measured using a Seca length meter.
Body Mass Index | at the 1st day
  Body weight and height will be combined to report body mass index in kilogram per meter squared.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Vrije Universiteit Brussel, Brussels
  - KU Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No
The Investigator and the Participating Site shall treat all information and data relating to the Study disclosed to Participating Site and/or Investigator in this Study as confidential and shall not disclose such information to any third parties or use such information for any purpose other than the performance of the Study. The collection, processing and disclosure of personal data, such as patient health and medical information is subject to compliance with applicable personal data protection and the processing of personal data (Directive 95/46/EC and Belgian law of December 8, 1992 on the Protection of the Privacy in relation to the Processing of Personal Data).
  Data are anonymous if no one, not even the researcher, can connect the data to the individual who provided it. No identifying information is collected from the individual.